CLINICAL TRIAL: NCT02547532
Title: Microbioma in Sputa From COPD With Alpha-1 Antitrypsin Deficiency
Acronym: AATD
Status: Completed | Type: Observational
Sponsor: Fondazione Salvatore Maugeri (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Bruno Balbi, Head, Pulmonary Rehabilitation Department, Fondazione Salvatore Maugeri
Other Study IDs: Fsalvatoremaugeri
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: COPD; alpha-1 antitrypsin deficiency; microbioma
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- usual COPD: Patients meeting the diagnostic criteria for COPD and without AATD
  Interventions: Other: collection of sputum
- normal smokers: subjects with a history of smoking, without symptoms, without AATD and with normal lung function
  Interventions: Other: collection of sputum
- normal non smokers: subjects without a history of smoking, without symptoms, without AATD and with normal lung function
  Interventions: Other: collection of sputum
- AATD not treated: patients with COPD, with AATD and not on augmentation therapy for AATD
  Interventions: Other: collection of sputum
- AATD treated: patients with COPD, with AATD on augmentation therapy for AATD
  Interventions: Other: collection of sputum

INTERVENTIONS:
Other: collection of sputum

SUMMARY:
In the context of the increasing evidence of the pathogenetic role of microbiome in COPD, our aim is to determine the total and specific bacterial and viral load in sputa from patients with COPD due to AATD and to correlate these findings with cellular, biochemical and immunological characteristics of sputa. These quantitative data obtained from sputum will be analyzed in the context of the clinical and physiological parameters of the patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD and a clinical stable condition, i.e. at least three months from the last AECOPD and/or antibiotic treatment.

For patients with AATD this condition will be diagnosed by laboratory tests showing low levels of AAT and genotyping of AATD-related genes.

. Exclusion Criteria:

* The presence of important co-morbidities (diabetes, systemic or organ infections, immunodeficiency, tumors, moderate-severe heart failure) will be considered as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunterrs Patients with COPD without AATD Patients with COPD and with AATD
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
composition of microbioma in sputa | 2 years

SECONDARY OUTCOMES:
correlation with clinical and physiological parameters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pantaleo Giannuzzi, M.D., Study Director — Fondazione Salvatore Maugeri